CLINICAL TRIAL: NCT00946374
Title: A Prospective Phase II Trial on R-CHOP Followed by High-dose BEAM and Autologous SCT and HLA-identical Allogenic SCT After Dose-reduced Conditioning in Patients Age < 55 Years With Primary Mantle-Cell-Lymphoma
Brief Title: Prospective Trial on Immunochemotherapy Plus Autologous Stem Cell Transplantation (SCT) and Allogenic SCT in Primary Mantle-Cell-Lymphoma
Acronym: HD-MCL2003
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Dr. med. A. D. Ho, University of Heidelberg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-149/2003; BfArM: A-7140-00-37/4021157
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2009-07-27 (Estimated); Status verified 2009-07

CONDITIONS: Mantle-Cell Lymphoma
Keywords: Mantle-Cell-Lymphoma; MCL; Non Hodgkin´s Lymphoma; NHL; Immunochemotherapy; R-CHOP; CHOP; High-dose chemotherapy; BEAM; HD-BEAM; Autologous stem cell transplantation; Reduced conditioning regimen; Unrelated donor; Sibling donor; Total Body Irradiation; TBI; Allogenic stem cell transplantation; ABSCT; ASCT; Fludarabine+TBI
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — R-CHOP protocol; Rituximab; Cyclophosphamide; Vincristine; Doxorubicin; Prednisone; Adrenal Cortex Hormones; Steroids; liposomal doxorubicin; Carmustine; Cytarabine; Etoposide; etoposide phosphate; Melphalan; Transplantation Conditioning; fludarabine phosphate; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Immunochemotherapy — R-CHOP: Rituximab 375 mg/m²,intravenous ( iv ), day 0 ; Cyclophosphamide 750 mg/m²,iv, day1; Vincristine 1,4 mg/m² but at the maximum 2 mg,iv,d1; Doxorubicin 50 mg/m², iv, d1; Prednisone 100 mg, peroral ( po ), day 1 to day 5
  Other Names: R-CHOP; CHOP; MabThera®; Endoxan®; Cytoxan®; Neosar®; Procytox®; Revimmune®; Oncovin®; Adriamycin®; Decortin®; Corticosteroid; Steroid; Cellcristin®; CAELYX®; Adriblastin®; Doxo-Cell®
Drug: High-dose BEAM plus autologous SCT — High-dose BEAM: Carmustine 300mg/m², iv, day -7; Cytarabine 2 x 200 mg/m², iv, day -6 to day -3; Etoposide 2 x 100 mg/m², iv, day -6 to day -3; Melphalan 140 mg/m², iv, day -2 followed by Autologous stem cell transplantation ( > 2,5 x 10e6 CD34 positive autologous stem cells, iv, day 0
  Other Names: BEAM; High-dose BEAM; ABSCT; ASCT; BCNU; Crmubris®; ARA-C; Eposin®; Etopophos®; ETO CELL®; Vepesid®; VP-16®; Alkeran®
Other: HLA-identical allogenic SCT — Fludarabine 30 mg/m², iv, day -4 to day -2; Cyclosporin A 2 x 3mg/kg, iv, day -1 to day 0 plus total body irradiation with 2 Gy, day 0 followed by allogenic stem cell transplantation immediately after Radiation.
  Other Names: Sibling donor; Unrelated donor; HLA-identical; Conditioning regimen; Fludara®; Sandimmune®; Fludarabinphosphat; Neoflubin®; TBI; Ciclral®

SUMMARY:
The purpose of this study is to improve the overall survival of Mantle-Cell-Lymphoma (MCL) by a new concept of treatment with primary curative intention consisting of six courses of immunochemotherapy followed by high-dose chemotherapy and autologous stem cell transplantation (SCT) and HLA-identical allogenic SCT after a dose-reduced conditioning regimen of total body irradiation (TBI) with 2 Gy and Fludarabine in younger patients with primary Mantle-Cell-Lymphoma

DETAILED DESCRIPTION:
With a median overall survival of approximately 3 years, MCL has the poorest prognosis of all NHL entities. No potentially curative therapy has been established yet as even more intensive therapies including high-dose chemotherapy plus autologous SCT show only moderate improvement of the prognosis of MCL. Allogenic SCT seems to have an immunological mechanism of action in NHL, which is commonly known as Graft-versus-Lymphoma effect. This trial´s purpose is to improve the overall survival in patients younger than 55 years with primary MCL by sequentially combining autologous SCT and allogenic SCT after the application of 6 courses of immunochemotherapy and high-dose chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. First diagnosis of Mantle-Cell-Lymphoma without any previous therapies except for pre-phase treatment consisting of steroids
2. Age 18 to 55 years
3. Confirmed CD20-expression on lymphocytes
4. Effective methods of contraception and negative pregnancy test
5. Sufficient compliance
6. Written patient´s informed consent

Exclusion Criteria:

1. Manifest cardiac insufficiency, not compensated
2. Congestive Cardiomyopathy
3. Chronic pulmonary disease including hypoxemia
4. Severe hypertension, not condensable with drugs
5. Severe diabetes mellitus not condensable with drugs
6. Renal Insufficiency ( serum creatinin > 2,0 mg/dl, other than Lymphoma related)
7. Liver impairment ( Transaminases value more than 3 x upper normal value or Bilirubin > 2,0 mg/dl, other than Lymphoma related)
8. HIV-Infection
9. Active Hepatitis B-Infection if continuous virostatic treatment is not possible
10. Active Hepatitis C-Infection
11. Clinical signs of cerebrovascular insufficiency or cerebral damages
12. Pregnancy, lactation or inadequate contraception in women of childbearing age
13. Severe psychiatric disorders
14. Transplantation in the past

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-07; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy: ORR, OS, EFS | during treatment and on day 720 after allogenic SCT

SECONDARY OUTCOMES:
Toxicity according to WHO-Grading | During treatment and until follow-up
GvL-effect after allogenic SCT | Allogenic SCT until day 720 after transplantation
Comparison of OS between patients completing the protocol and patients not receiving allogenic SCT | First diagnosis of MCL until day 720 after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D. Ho, Ph.D., Prof., Principal Investigator — Director of Department
Locations (1):
- University Hospital, Heidelberg, Germany

REFERENCES:
- See also: Homepage University hospital Heidelberg, Germany — http://www.klinikum.uni-heidelberg.de